CLINICAL TRIAL: NCT05594459
Title: Early Treatment With Invasive Technique in Cancer Pain Management, Impact on Patient's Quality of Life. A Randomized Clinical Trial
Brief Title: Early Treatment With Invasive Technique in Cancer Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, MD, Director of Anesthesiology and Intensive Care Utin, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: V1.18.10.22
Record Dates: First submitted 2022-10-19; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cancer Pain; Opioid Use
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioids (Active Comparator)
  Interventions: Drug: high opioids dosages
- Mini invasive (Experimental)
  Interventions: Procedure: Mini invasive analgesic technique

INTERVENTIONS:
Procedure: Mini invasive analgesic technique — patients will be treated with early interventional neuromodulatory techniques, before high opioids dosages.
  Arms: Mini invasive
Drug: high opioids dosages — patients will be treated with high opioids dosages
  Arms: Opioids

SUMMARY:
Background: high or moderate intensity pain hits more than a half of patients with cancer and is not adequately treated way in 1/3 of this patients. Complexity of cancer pain makes right management difficult and the consequences of an incorrect management are far-reaching in a clinical and social way. A multimodal treatment tailored on the patient, and the evaluation of quality of life correlated to different treatment methodologies, must constitute a decisive element in terms of therapeutic choices.

Over the past 30 years, the World Health Organization (WHO) analgesic step ladder has been used to guide the choices management of cancer-related pain, but in the last years the growth of innovative treatment strategies, led to the need to modulate this rigid yet useful system. Benefits would be obtained with interventional techniques (peripheral neural blockade, neuromodulatory device use, neuro-destructive techniques, and intrathecal drug delivery systems) performed in the initial parts of the treatment cycle (before the third step of the WHO scale), rather than applied according to the WHO scale algorithm. Some authors who adopted this approach, reported reduction in pain duration and less opioid consumption, minimizing the risk of opioid related side effects and an improving the overall quality of life .

The hypothesis is that early application of interventional techniques in oncological patients has an improving effect in the treatment of chronic cancer pain in terms of efficacy and quality of life.

Materials and methods: patients followed by the Cancer Pain Therapy Service of the Cancer National Institute Regina Elena, Rome, with chronic localizable abdominal pain with a value ≥ 7 according to the numeric rating scale (NRS) and a diagnosis of untreatable disease will be randomized into two groups: in the first group patients will be treated with early interventional neuromodulatory techniques, before high opioids dosages. The other group will follow the steps of the WHO scale.

Every patient will receive the European Organization for Research and Treatment of Cancer Quality of life-Core 30 Summary Score (EORTC-QLQ C30) survey to detect quality of life and the Numeric rate scale NRS. They will receive it before the treatment, after invasive procedure, one month later and six months later.

Primary end point will be the difference of the quality of life questionnaire score between the groups; secondary end point will be difference in the NRS values. The statistic analysis will be based on two groups of patients responding to the including criteria. The sample will be made of 76 patients divided in two sub-sample of equal dimension to select and analyze in 18 months. The sample thus defined is consistent for a confidence interval of 80% and for a margin of error of less than 5%.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an oncological disease defined as not curable
* Pain localized in the abdomen, described as severe with NRS ≥ 7
* American Society of Anesthesiology status ≤ III
* Karnofsky performance status scale ≥60%
* Written informed consent

Exclusion Criteria:

* Inability to answer / fill in questionnaires
* Patients under psychotherapy treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-11-25 (Estimated); Primary Completion 2024-07-25 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in European Organization for Research and Treatment of Cancer Quality of life-Core 30 Summary Score (EORTC-QLQ C30) | V0 (up to 2 weeks), V1 (One month after), V2 (3 months later)
  difference of the quality of life questionnaire score between the groups

IPD SHARING:
Plan to Share IPD: No